CLINICAL TRIAL: NCT01771029
Title: Technical Evaluation of a Whole Blood Rapid Test Measuring Procalcitonin (BRAHMS PCT Direct)
Brief Title: Technical Evaluation of Brahms PCT Direct
Status: Completed | Type: Observational
Sponsor: Philipp Schuetz (Other)
Collaborators: Thermo Fisher Scientific, Inc (Industry)
Responsible Party: Sponsor-Investigator, Philipp Schuetz, PD Dr. med. Oberarzt, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Other Study IDs: POC_1
Record Dates: First submitted 2013-01-09; First posted 2013-01-18 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Infection
Keywords: Procalcitonin; Infection; Point-of-Care
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Validation of the technical performance of the BRAHMS PTC direct point-of-care assay under routine conditions with native patient samples. The clinical validation is planned as a method comparison to a reference method (BRAHMS PCT sensitive KRYPTOR, Elecsys BRAHMS PCT). The study hypothesis is to show a highest correlation between the new product and the reference methods.

DETAILED DESCRIPTION:
Procalcitonin (PCT) is a highly sensitive and specific marker which can be detected in the blood stream in response to a bacterial infection. In contrast to conventional infection disease markers PCT permits the differential diagnosis between bacterial and viral infections. The marker is implemented on Intensive Care Units (ICU) and Emergency Departments (ED) worldwide since 1996. Until now various technologies all basing on the use of serum or plasma samples are available in the market.

BRAHMS GmbH (Clinical Diagnostics Division of Thermo Fisher Scientific) as manufacturer of the Procalcitonin assays has developed a new quantitative immunochromatographic whole blood point-of-care assay, the BRAHMS PCT direct. The test follows the principle of a sandwich assay with two anti-PCT antibodies, one immobilized on a nitrocellulose membrane and the tracer antibodies labeled with gold.

Validation of the technical performance of the product under routine conditions with native patient samples. The clinical validation is planned as a method comparison to a reference method (BRAHMS PCT sensitive KRYPTOR, Elecsys BRAHMS PCT). The internal pre-studies were performed with blood samples spiked with recombinant PCT and with native patient samples.

The primary objective of this study is to show a highest correlation between BRAHMS PCT direct with the PCT reference method for PCT- positive and negative samples.

The secondary object of this study is to show the advantage of BRAHMS PCT direct in time to result in comparison to the reference method.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* possible infection at initial presentation
* informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One cohort of 150-250 patients, possible infection at initial presentation in Kantonsspital Aarau.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2013-02; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Correlation between BRAHMS PCT direct and reference method. | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Showing at least 90% correlation between BRAHMS PCT direct with the PCT reference method for PCT- positive and negative samples.

SECONDARY OUTCOMES:
Time to result | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  The secondary object of this study is to show the advantage of BRAHMS PCT direct in time to result in comparison to the reference method.

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Schuetz, PD, Dr.med., Principal Investigator — Kantonsspital Aarau
Locations (3):
- Pitié Salpetrière. Groupement hospitalière universitaire Est, Paris, Paris, France
- Klinikum Ernst von Bergmann, gemeinnützige GmbH Akademisches Lehrkrankenhaus der Humboldt-Universität Berlin (Charité), Potsdam, Germany
- Kantonsspital Aarau Innere Medizin, Aarau, Canton of Aargau, Switzerland